CLINICAL TRIAL: NCT05752877
Title: Clinical Study on Evaluation of Safety and Efficacy of Targeted IL-13 Rα2 or B7-H3 UCAR-T Cell Injection in Treatment of Advanced Glioma
Brief Title: Safety and Efficacy of Targeted IL-13 Rα2 or B7-H3 UCAR-T for Advanced Glioma
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital of Soochow University (Other)
Collaborators: Soochow T-Maximun Biotechnology Co. LTD (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SJWKtumor001
Record Dates: First submitted 2023-02-20; First posted 2023-03-03 (Actual); Last update posted 2023-03-03 (Actual); Status verified 2023-02

CONDITIONS: Advanced Glioma; Complication of Chimeric Antigen Receptor (CAR-T) Cell Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Interventional Group (Experimental)
  Interventions: Biological: Targeted IL-13 Rα2 UCAR-T cell injection; Biological: Targeted B7-H3 UCAR-T cell injection

INTERVENTIONS:
Biological: Targeted IL-13 Rα2 UCAR-T cell injection — local administration (intracranial cavity or intravertebral injection after surgery): 1 ampoule (about 2-5 ml, 1-5×10^7 cells) for 1-2 minutes each time.
Biological: Targeted B7-H3 UCAR-T cell injection — local administration (intracranial cavity or intravertebral injection after surgery): 1 ampoule (about 2-5 ml, 1-5×10^7 cells) for 1-2 minutes each time.

SUMMARY:
The goal of this clinical trial is to estimate the safety, tolerance and initial efficacy of target IL-13Rα2 or B7-H3 UCAR-T cell injection in the treatment of patients with advanced glioma, as well as the pharmacokinetic characteristics of its metabolites after single and multiple administrations and the biomarkers related to efficacy, safety and drug metabolism.

ELIGIBILITY:
Inclusion Criteria:

* 18-70 years old, male or female, and the expected survival period is not less than 3 months.
* Advanced, locally advanced or recurrent tumor diagnosed histologically or cytologically.
* Failed in previous standard treatment or gived up treatment for various reasons after failure of first-line treatment.
* Failed in therapy by PD-1 or PD-L1 antibody or stopped administration of PD-1 or PD-L1 antibody for more than 4 weeks.
* At least 1 measurable target lesion (RECIST v1.1).
* 0-2 in ECOG physical state score.
* Available initial or recurrent tumor tissue for at least 10 stanable and detectable sections.
* Blood routine test: WBC ≥ 3×10^9/L, lymphocyte percentage (LY%) ≥ 15%, hemoglobin Hbo (Hb) ≥ 90g/L, platelet (PLT) ≥ 60×10^9/L.
* Liver and kidney functions: alanine transaminase (ALT) and aspartate transaminase (AST) < 3 times of the normal value, total bilirubin (TBiL) < 1.5 times of the normal value, serum creatinine (SCR) < 1.5 times of the normal value.
* IL-13Rα2 or B7-H3 antigen expression > 50%.
* Volunteered to enroll this study and signed the informed consent with good compliance and cooperation with follow-up.
* Experienced radiotherapy and chemotherapy with an interval of more than 4 week.

Exclusion Criteria:

* Hepatitis B surface antigen (HBsAg) or hepatitis B core antibody (HBcAb) positive and peripheral blood HBV DNA titer ≥ 5 × 10^2 copies/L; HCV antibody and peripheral blood HCV RNA positive; Human immunodeficiency virus (HIV) antibody positive; CMV DNA test positive; Syphilis test positive.
* Experienced any gene therapy previously.
* Needing long-term immunosuppressants for any reason.
* Any serious and uncontrolled systemic autoimmune disease or any unstable systemic disease, including but not limited to systemic lupus erythematosus, rheumatoid arthritis, ulcerative colitis, Crohn's disease and temporal arteritis.
* Severe heart, lung, liver and kidney insufficiency or severe debilitating lung disease; Cardiac function: Grade III or above according to NYHA standard; Liver function: grade C in Child-Puge grading standard; Renal function: chronic kidney disease (CKD) more than stage 4; Renal insufficiency above stage Ⅲ; Lung function: symptoms of severe respiratory failure, involving other organs; Brain function: abnormality of central nervous system or disturbance of consciousness.
* Administrating of systematical steroids currently (except usage inhaled steroids recently or currently).
* Pregnancy and lactation (the safety of this treatment for unborn children is not clear, and female participants with reproductive potential must have negative serum or urine pregnancy test within 48 hours before administration).
* Allergy to immunotherapy and related drugs.
* Complicated with another tumor.
* History of organ transplantation or waiting for organ transplantation.
* After evaluation by researcher,noncompliance with the requirements of the study protocol was confirmed.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2021-05-01 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate | Up to 5 years or complete the follow-up of the last enrolled patient, whichever comes first.
  The proportion of patients whose tumor size decreases to the expected value and can continue to meet the expected minimum time limit。

SECONDARY OUTCOMES:
Progression-Free Survival | Up to 5 years or complete the follow-up of the last enrolled patient, whichever comes first.
  The time from enrolling into the trial to the first occurrence of disease progression or death from any cause。

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China